CLINICAL TRIAL: NCT04881253
Title: COVID-19 Patient Cohort: Retinal Damage in Non-invasive Retinal Imaging (OCTA)
Status: Terminated | Type: Observational
Why Stopped: End of covid crisis
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-RET
Record Dates: First submitted 2020-11-02; First posted 2021-05-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Covid19; Retina Injury
Keywords: OCT-A; OCT
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this research is to build a collection of non-invasive retinal imaging (OCT and OCTA) in order to investigate the incidence and impact of retinal damage in patients who have or have had COVID-19.

DETAILED DESCRIPTION:
This monocentric study is aimed at 3 types of patients:

* Those who have been hospitalized for Covid-19 during the epidemic
* Newly infected and diagnosed patients Covid-19
* Those with paucisymptomatic Covid-19 who did not require hospitalisation

At the patient's inclusion, an ophthalmologic assessment will be performed including :

* visual acuity,
* SD-OCT + multicolor,
* OCT-A,
* color retinography,

Fundus examination, optical coherence tomography (OCT) and optical coherence tomography angiography (OCTA) in all COVID-19 patients may detect retinal lesions. In addition, if a correlation is demonstrated between clinical and paraclinical parameters and between disease severity and retinal vascular damage in non-invasive imaging (OCT and OCTA), this would allow a better understanding of the pathophysiology of the disease, as well as factors that may influence disease severity and the mechanisms potentially responsible for the observed disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Diagnosis of COVID-19 proven on RT-PCR, antigenic test or chest CT scan
* Affiliation to the general social security system
* A consent signed by the patient

Exclusion Criteria:

- Refusal of patient participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with COVID-19, patients who were hospitalised for COVID-19 and patients with COVID-19 who did not require hospitalisation
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Retinal damage at inclusion after Covid-19 infection | Up to one week after inclusion
  Comparison of retinal damage in patients with patients with severe forms of Covid-19 versus patients with mild forms of the disease

SECONDARY OUTCOMES:
Change of retinal vascular density at inclusion after Covid-19 infection | Up to one week after inclusion
  Comparison of retinal damage in patients with severe forms of Covid-19 versus patients with mild forms of the disease
Impact of retinal vascular density changes on visual acuity at inclusion | Up to one week after inclusion
  Severity and impact of retinal damage
Presence of Retinal toxicity (atrophy) on multimodal retinal imagery | Up to one week after inclusion
  Correlation between the presence of changes in multimodal imaging (fundus autofluorescence, multicolor and OCTA) and the associated antiviral treatment for Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, IDF, France

IPD SHARING:
Plan to Share IPD: No